CLINICAL TRIAL: NCT05746325
Title: Pilot Feasibility Study of Tumor Treating Fields in Treatment of Leptomeningeal Metastases Involving the Spine
Brief Title: Tumor Treating Fields for the Treatment of Leptomeningeal Metastases of the Spine in Patients With Breast or Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210303; NCI-2023-00240 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-005732 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-02-14; First posted 2023-02-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Leptomeninges; Metastatic Lung Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis; Lung Neoplasms | interventions — Spinal Puncture; Magnetic Resonance Spectroscopy; Physical Examination; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (TTFields, digital photos) (Experimental): Patients have transducer arrays applied and digital photographs taken of placement on study. Patients wear the NovoTTF-200T portable system on study. Patients also undergo MRI and may undergo LP during screening and on study.
  Interventions: Other: Digital Photography; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Device: Medical Device Usage and Evaluation; Procedure: Biospecimen Collection

INTERVENTIONS:
Other: Digital Photography — Digital photographs taken of array placement
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Device: Medical Device Usage and Evaluation — Transducer arrays applied and wear NovoTTF-200T
Procedure: Biospecimen Collection — Undergo collection of cerebrospinal fluid (CSF) during screening if no CSF testing for malignancy has been done previously
  Other Names: Biological Sample Collection; Specimen Collection

SUMMARY:
This clinical trial evaluates the safety and feasibility of tumor treating fields (TTF) in the treatment of spinal leptomeningeal disease in patients with breast or lung cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Patients wear the portable Novo TTF-200T device that produces electric fields to target areas on the body to stop the growth of tumor cells. The information from this study will help researchers develop a better treatment for leptomeningeal metastases in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the TTF device can be successfully placed in the three protocol-specified treatment field arrays (cervical, thoracic, and lumbar) and worn by the study patients for a meaningful period of time in the treatment of leptomeningeal metastases within the spine.

SECONDARY OBJECTIVE:

I. To document any preliminary signals of activity, as measured by radiographic and clinical response, or durable stability of objective neurologic examination, utilizing Leptomeningeal Assessment in Neuro-Oncology (LANO) criteria, magnetic resonance imaging (MRI) imaging, cerebrospinal fluid (CSF) cytologic examination, and patient-reported symptom assessment (M. D. Anderson Symptom Inventory [MDASI]-spine module).

OUTLINE:

Patients have transducer arrays applied and digital photographs taken of placement on study. Patients wear the NovoTTF-200T portable system on study. Patients also undergo MRI during screening and on study and may undergo lumbar puncture (LP) and collection of cerebrospinal fluid (CSF) samples during screening if no CSF testing for malignancy has been done previously.

After completion of study intervention, patients are followed up every 3 months or every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Prior tissue diagnosis of breast cancer or lung cancer
* Confirmed diagnosis of leptomeningeal metastases (LM) with positive cerebrospinal fluid (CSF) cytology for malignancy and meningeal enhancement (type 1A, 1B, and 1C)
* Radiographic evidence on MRI of leptomeningeal enhancement within the cervical, thoracic or lumbar spine on spinal MRI
* Life expectancy of at least 6 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2, or 3
* Recovery from any neurotoxic effects of prior therapy
* Platelet count greater than 25 x 10^9/L
* Absolute neutrophil count (ANC) greater than 0.5 x 10^9/L
* Patients must have adequate liver function, total bilirubin < 2.5 mg/dL, unless elevated total bilirubin is due to elevated indirect bilirubin from known Gilbert's disease, aspartate aminotransferase (AST) =< 3.5 times upper limits of normal; adequate renal function [calculated estimated glomerular filtration rate (eGFR) >= 30 mL/min/ body surface area (BSA)]
* Patients or legal medical representative must provide written informed consent
* Patients must have suitable body habitus for placement of transducer arrays
* Patients must be willing to wear the device for at least 18 hours a day (averaged over monthly)
* Patients must be willing to return for the scheduled evaluations and perform the required assessments
* Patients are without other disease or situation which would significantly compromise adequate assessment of safety and feasibility of the TTF
* Patient willing to start a study treatment with TTF =< 14 days from registration

Exclusion Criteria:

* Concomitant therapy:

  * Must not be receiving concurrent high-dose methotrexate (>= 3 g/m^2), high dose thiotepa, or high-dose cytarabine (>= 3 g/m^2). Any other systemic chemotherapy, targeted treatment, hormonal or immunotherapy directed at the primary systemic malignancy is permitted
  * Must not have received radiation therapy (RT) to the brain or spinal cord within 2 weeks of initiation of TTF
  * Must be at least 1 week from cessation of any prior intrathecal chemotherapy
* Women of childbearing age who are pregnant or lactating. (Male and female patients who are fertile must be willing to use an effective means of birth control to avoid pregnancy)
* Patients with uncontrolled or untreated infection including active hepatitis, and human immunodeficiency virus (HIV)
* Patients receiving any other investigational agents and must not have received any other investigational agent within 14 days prior to registration. The 14-day period should be extended if the investigational agent is known to have delayed toxicity
* Patients known to be allergic to the hydrophilic gel utilized for transducer attachment
* Patients with surgical hardware within the planned area of treatment in the spine (e.g., titanium rods, screws, fixation devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of significant toxicity of tumor treating fields (TTFs) | Up to 3 years
  Will be measured by incidence of grade 3 or greater non-hematologic adverse events that persist despite temporary interruption of treatment and maximal medical management (i.e., grade 3 or greater non-hematologic toxicities that are not responsive to cessation of treatment and administration of supportive care). Toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Feasibility of TTFs - completion of at least 28 days of TTF therapy | Up to 28 days
  Assessed by the number of patients who are unable to complete at least 28 days of TTF therapy (a composite average for the 28 days of at least 50% of array 'on' time) due to unacceptable adverse events. Treatment with TTF will be considered feasible if the stopping rule is not reached, as defined per protocol.

SECONDARY OUTCOMES:
Preliminary signals of activity - CSF cytologic response | Up to 3 years
  Descriptive analyses will be performed to assess preliminary signals of activity. CSF cytologic response will be assessed for patients who had positive CSF cytology at baseline.
Preliminary signals of activity - MRI radiographic response | Up to 3 years
  Descriptive analyses will be performed. Assessed by MRI radiographic response within the TTF field
Preliminary signals of activity - time to CSF cytologic repsonse | Up to 3 years
  Descriptive analyses will be performed. Assessed by time to CSF cytologic response (patients with positive baseline CSF cytology only), defined as the date of initiation of TTF to the last date of three consecutive negative CSF cytologic examinations).
Preliminary signals of activity - duration of CSF cytologic response | Up to 3 years
  Descriptive analyses will be performed. Assessed by time from the date of the third consecutive negative CSF to CSF cytologic relapse (defined as either suspicious or positive cytology).
Preliminary signals of activity - neurologic progression-free survival | Up to 3 years
  Descriptive analyses will be performed. Assessed by neurologic progression-free survival, the time from study enrollment to documented worsening of neurological symptoms or signs of disease progression.
Preliminary signals of activity (defined as either suspicious or positive cytology). | Up to 3 years
  Descriptive analyses will be performed. Data evaluated will include: Duration of cytologic response (time from the date of the third consecutive negative CSF to CSF cytologic relapse (defined as either suspicious or positive cytology).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J. Sherman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials